CLINICAL TRIAL: NCT03222778
Title: Combination of Static Echocardiographic Indices for Prediction of Fluid Responsiveness During Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2017-0403
Record Dates: First submitted 2017-07-09; First posted 2017-07-19 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Fluid Responsiveness
Keywords: fluid responsiveness; tissue doppler; off-pump coronary bypass surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- hypovolemia (fluid responsiveness): The patients with fluid responsiveness (an increase in stroke volume index of ≥12%) after fluid challenge using 6 ml/kg of balanced 6% hydroxyethyl starch 130/0.4 (Volulyte; Fresenius Kabi, Bad Homburg, Germany)
- NO hypovolemia (NO fluid responsiveness): The patients without fluid responsiveness after fluid challenge using 6 ml/kg of balanced 6% hydroxyethyl starch 130/0.4 (Volulyte; Fresenius Kabi, Bad Homburg, Germany)

SUMMARY:
In the perioperative or critical care of hemodynamically unstable patients, appropriate fluid resuscitation guided by reliable preload indices is of pivotal importance as only half of them are fluid responsive, and that empiric fluid administration actually leads to dismal prognosis. In the continuum of being non-invasive, combinations of tissue Doppler-derived parameters of early (e') and late (a') diastolic, and peak systolic velocity (s') of the mitral annulus provide information regarding the systolic dysfunction and preload (e'/s'), and LV stiffness (e'/a'). Although the left ventricular end-diastolic area (LVEDA) alone is not a valid predictor of fluid responsiveness, combining LVEDA with these indices would provide comprehensive information regarding the LV dimension, preload, and compliance as well as systolic function. Also, it seems logical to assume that patients with low LVEDA and high e' velocity indicating preserved early diastolic relaxation or low e (early mitral inflow velocity) /e' ratio indicating normal LV filling pressure would more likely be fluid responsive. Yet, these assumptions have not been tested before. Moreover, these values can be reliably obtained regardless of the heart rhythm, except for a', and do not completely rely on heart-lung interaction as opposed to the dynamic indices. Thus, the aim of this prospective trial is to investigate the role of LVEDA combined with e, e', a' or s' as a preload index in predicting fluid responsiveness in patients scheduled for off-pump coronary bypass surgery, in closed-chest conditions.

ELIGIBILITY:
Inclusion Criteria:

1. the patients scheduled for off-pump coronary bypass surgery
2. tha age ≥20 yrs old
3. the patients who are willing to provide written informed consent

Exclusion Criteria:

heart rhythm other than sinus, L, septal and/or lateral wall motion abnormalities, and a

1. New York Heart Association functional class ≥III
2. LV ejection fraction <40%
3. emergency operation
4. the patients with preoperative septal and/or lateral wall motion abnormalities
5. contraindications to transesophageal echocardiography or balanced 6% hydroxyethyl starch 130/0.4
6. the patients with any valvular heart disease ≥moderate degree
7. No communication possible due to a language barrier or deafness

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients scheduled for off-pump coronary bypass surgery
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2020-03-06 (Actual)

PRIMARY OUTCOMES:
Predictive ability of combined echocardiographic index consisting of LVEDA, e, e', s' or a' | 15 to 20 min after anesthetic induction during closed chest condition
  Fluid challenge is performed once using 6 ml/kg of balanced 6% hydroxyethyl starch 130/0.4 (Volulyte; Fresenius Kabi, Bad Homburg, Germany) 15 to 20 min after anesthetic induction during closed chest condition. Fluid responsiveness is defined as an increase in stroke volume index of ≥ 15%. Assessment of echocardiographic variables [LVEDA, e, e', a' or s'] is performed before fluid challenge. We assess the predictive ability of a combined echocardiographic preload index consisting of LVEDA, e, e', s' or a' on fluid responsiveness using the area under the Receiver Operating Characteristic (ROC) curve (AUROC).

SECONDARY OUTCOMES:
Comparison between the combine echocardiographic index and LVEDA alone, CVP, PCWP, RVEDV and PPV for the predictive ability on fluid responsiveness | 15 to 20 min after anesthetic induction during closed chest condition
  CVP, PCWP, RVEDV and PPV are measured as well as echocardiographic variables [LVEDA, e, e', a' or s'] before fluid challenge. We also assess the predictive ability of LVEDA alone, CVP, PCWP, RVEDV and PPV on fluid responsiveness using each AUROC, and compare the predictive power of the combined echocardiographic index on fluid responsiveness with those of the LVEDA alone, CVP, PCWP, RVEDV, and PPV.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No